CLINICAL TRIAL: NCT05139862
Title: Neuro-cardiac Predictors of Treatment Response to RTMS in Depression: a Mechanistic Study Using Interleaved TMS-fMRI
Brief Title: Neurocardiac Predictors of Treatment Response to RTMS in Depression
Acronym: NCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, MD, PhD, FRCPC, DFAPA, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-00648
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Depression; Treatment Resistant Depression
Keywords: Repetitive Transcranial Magnetic Stimulation; rTMS; Neurostimulation; Heart Rate Variability; fMRI
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: For MDD patients, the study will consist of six weeks of rTMS treatment using intermittent theta burst stimulation (iTBS) rTMS to the left DLPFC. Treatment will be administered daily, 5 days per week (i.e., 30 treatments).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active iTBS (Experimental): Active intermittent theta-burst stimulation (iTBS) rTMS session on the left dorsolateral prefrontal cortex (L-DLPFC)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — This study utilizes intermittent theta burst stimulation (iTBS) to the left DLPFC.
  Other Names: rTMS

SUMMARY:
Heartbeat is controlled by the brain and is regular but flexible to change in response to environmental and internal stimuli. This feature is known as heart rate variability (HRV). Major depressive disorder (MDD) has been associated with diminished HRV and this is a reflection of abnormal brain function caused by MDD. Repetitive transcranial magnetic stimulation (rTMS) is a treatment that stimulates specific areas of the brain. The goal of this study is to test the hypothesis that rTMS induces changes in connectivity between the area of the brain stimulated with rTMS and deeper areas in the brain associated to heart rate regulation. 110 patients with TRD will be recruited and will undergo a concurrent TMS-fMRI session before receiving a course of iTBS to the L-DLPFC for 30 sessions at 120% rMT.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

1. are female or male;
2. are outpatients;
3. are voluntary and competent to consent to treatment;
4. have a DSM 5 diagnosis of MDD, single or recurrent confirmed by Mini-International Neuropsychiatric Interview (MINI) version 6.0;
5. are between the ages of 18 and 65 years;
6. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode OR have been unable to tolerate at least two separate trials of antidepressants at less than the minimum adequate dose and/or duration (ATHF 1 or 2);
7. A score ≥ 18 on the Hamilton Depression Rating Scale (HDRS-17 item);
8. Have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening;
9. Able to adhere to the treatment schedule;
10. pass the TMS and MRI adult safety screening questionnaires.

Exclusion Criteria:

Patients are excluded if they:

1. have a history of substance use within the last 3 months;
2. have a concomitant major unstable medical illness;
3. have active suicidal intent;
4. are pregnant;
5. have a lifetime (MINI) diagnosis of any psychotic or bipolar disorder;
6. have a MINI anxiety disorder or personality disorder assessed by a study investigator to be primary and causing greater impairment than MDD;
7. have ever failed a course of ECT;
8. have previously received rTMS;
9. have any significant neurological disorder, any history of seizure (except those therapeutically induced by ECT), significant head trauma with loss of consciousness for > 5 min;
10. have any intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
11. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to study entry, with no anticipated change in the frequency of therapeutic sessions, or focus of therapeutic sessions over the duration of the study;
12. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators;
13. are currently taking lorazepam greater than 2 mg daily (or equivalent) or any dose of an anticonvulsant, due to the potential to limit rTMS efficacy;
14. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview);
15. have failed more than three adequate trials (ATHF > 3) of medication in the current episode.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Depressive Symptoms using HDRS-17 Scale at Week 10 | Baseline and Week 10
  The 17-item Hamilton Depression Rating Scale (HRSD-17) will be used as the primary outcome measure as well as the tool to establish severity cut off for eligibility (Hamilton, 1960). The scoring ranges from 0-52, with higher scores indicating more severe depression symptoms.

SECONDARY OUTCOMES:
Change from Baseline in Anxiety Symptoms using HAM-A Scale at Week 10 | Baseline and Week 10
  The 14-item Hamilton Anxiety Rating Scale (HAM-A) will be used as a secondary outcome measure in this study. The scoring of this assessment ranges from 0-56, with higher scores indicating more severe anxiety symptoms.
Change from Baseline in Depressive Symptoms using QIDS-16 Scale at Week 10 | Baseline and Week 10
  The self-rated 16-item Quick Inventory of Depressive Symptoms (QIDS-16) will be used as a secondary outcome measure in this study. The scoring of this assessment ranges from 0-27, with higher scores indicating more severe depression symptoms.

OTHER OUTCOMES:
Change from baseline in Heart Rate Variability at Week 10 | Baseline and Week 10
  Heart Rate Variability metrics

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, M.D., Ph.D., Principal Investigator — Department of Psychiatry, UBC
Locations (1):
- Non-Invasive Neurostimulation Therapies (NINET) Laboratory, UBC Department of Psychiatry, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No